CLINICAL TRIAL: NCT06589453
Title: Evaluation of Nasal Elevator Versus Grayson's Nasal Stent in Conjunction with Digital Nasoalveolar Molding (D-NAM) Appliance on Nasolabial Esthetics in Infants with Bilateral Cleft Lip and Palate: a Randomized Clinical Trial
Brief Title: Evaluation of Nasal Elevator Versus Grayson's Nasal Stent with D-NAM Appliance on Nasolabial Esthetics in Bilateral Cleft Lip and Palate Infants
Acronym: D-NAM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, : Donia Ayman Ahmed Ezzeldin ElSayed, Assistant lecturer at Orthodontic Department, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-NAM 2024
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Cleft Lip and Cleft Palate
Keywords: Cleft lip and palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasal stent with Digital Nasoalveolar molding (Active Comparator)
  Interventions: Device: Nasal stent with digital nasoalveolar molding in bilateral cleft lip and palate infants
- Nasal elevator with Digital Nasoalveolar molding (Experimental): Nasal elevator will be used in conjunction with digital nasoalveolar molding appliance to improve nasolabial esthetics in bilateral cleft lip and palate infants.
  Interventions: Device: Nasal elevator with digital nasoalveolar molding in bilateral cleft lip and palate infants

INTERVENTIONS:
Device: Nasal elevator with digital nasoalveolar molding in bilateral cleft lip and palate infants — This is a unique nasal elevator aiming to improve nasolabial esthetics in conjunction with digital nasoalveolar molding appliance when used in bilateral cleft lip and palate infants.
  Arms: Nasal elevator with Digital Nasoalveolar molding
Device: Nasal stent with digital nasoalveolar molding in bilateral cleft lip and palate infants — Nasal stent that is used in conjunction with digital nasoalveolar molding in bilateral cleft lip and palate infants
  Arms: Nasal stent with Digital Nasoalveolar molding

SUMMARY:
Newborns with bilateral cleft lip/ palate will be treated pre-surgically by either nasal elevator or Grayson nasal stent in conjunction with digital nasoalveolar molding (D-NAM) appliance in order to evaluate their effect on the nasolabial esthetics.

DETAILED DESCRIPTION:
The aim of this trial is to evaluate and compare the short-term effect of nasal elevator with Grayson nasal stent in conjunction with digital nasoalveolar molding appliances at 2 stages T1 (Before NAM therapy), and T2 (After NAM therapy) as regards nasolabial esthetics and maxillary arch changes.

Newborns with Bilateral cleft lip/ palate will be allocated randomly into two groups: the first group will receive nasal elevator with digital nasoalveolar molding appliance while the second group will receive Grayson nasal stent with digital nasoalveolar molding appliance. The follow-up period will be 4-6 months till surgical lip closure. The nasolabial esthetics will be assessed using facial scans and 2D photographs, while changes in the maxillary arch will be assessed by digital maxillary models.

ELIGIBILITY:
Inclusion Criteria:

* Non-syndromic Infants with complete BCLP infants
* Infants less than 1 month of age.
* Males and females.
* Infants with displaced premaxilla
* Patients whose parents provided written consent for the study.

Exclusion Criteria:

* Patients above 1 month of age.
* Syndromic and systemically ill infants.
* Patients with unilateral cleft lip and palate.
* Incomplete Cleft lip or Simonart band (soft tissue bridge at the cleft side).
* Medically compromised patients
* Patien parents/guardians who will be unwilling to go through the Naso-alveolar molding (NAM) therapy.

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Nasolabial esthetics | 4-6 months
  Columellar length is to be measured in millimeters digitally using facial scans before and after Nasoalveolar Molding therapy.

SECONDARY OUTCOMES:
Maxillary arch changes | 4-6 months
  Maxillary arch changes will be assessed in millimeters using maxillary digital models.

IPD SHARING:
Plan to Share IPD: Undecided